CLINICAL TRIAL: NCT01654848
Title: Heparin-induced Thrombocytopenia (HIT II) in Liver Transplant Recipients: a Prospective Multivariate Analysis of Prognostic Factors and Haemostaseological Findings
Brief Title: Heparin-induced Thrombocytopenia (HIT II) in Liver Transplant Recipients
Acronym: HITOLT
Status: Completed | Type: Observational
Sponsor: CHIR-Net (Network)
Collaborators: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: TransplanTUM-1; HITafterOLT (Other: TransplanTUM)
Record Dates: First submitted 2012-03-30; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Heparin-induced Thrombocytopenia; Liver Transplantation
Keywords: liver transplantation; thrombocytes; heparin-induced thrombocytopenia; multivariate analysis of associated factors of HIT 2 after OLT; laboratory investigations of HIT-antibodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- orthotopic Liver Transplantation: consecutive inclusion of all recipients

SUMMARY:
In a prospective observational study the incidence of Heparin-induced Thrombocytopenia (HIT) Type 2 after orthotopic liver transplantation, associated factors, and hemostaseological findings in thrombocytes and anti-body patterns is going to be investigated.

DETAILED DESCRIPTION:
The investigators examined the frequency of anti-PF4/heparin antibodies (IgG/M/A; EIA) and their functional activity (HIPA) in 38 whole organ deceased donor liver transplant recipients. Additionally, demographic, clinical, donor- and recipient-specific parameters and laboratory findings (ALAT, ASAT, cholinesterase) were investigated.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive liver transplant recipients between 01/2010 and 08/2011 who
* were transplanted at our center after allocation of a liver graft via Eurotransplant

Exclusion Criteria:

* patient's refusal to participate in prospective observation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive livertransplant recipients of our transplant center, organ allocation via Eurotransplant Foundation, Leiden, The Netherlands; Laboratory investigations performed at the Abteilung für Transfusionsmedizin am Institut für Immunologie und Transfusionsmedizin der Universitätsmedizin Greifswald, Greifswald, Germany
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Assfalg, MD, Principal Investigator — Klinikum rechts der Isar, Dept. of Surgery
Locations (1):
- Klinikum rechts der Isar der TU München, Munich, Germany